CLINICAL TRIAL: NCT06530589
Title: Effects of Tupler's Technique on the Management of Diastasis Rectus Abdominis in Post-Partum Females.
Brief Title: Effects of Tupler's Technique on the Management of Diastasis Rectus Abdominis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Aqsa Shahid
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Diastasis Rectus Abdominis
Keywords: Diastasis Rectus Abdominis; Post-Partum Period; Tupler's Technique; Abdominal Strength

STUDY DESIGN:
Intervention Model Description: There will be comparison between two groups, experimental and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Tupler's Technique will be applied to this group. This technique includes Tupler's technique exercises and patients will also wears diastasis rehab splints. Patients will perform seated isometric exercises (elevator and contracting exercises) after wearing diastasis rehab splint. Repetitions of exercises will be 100 and whole intervention will be provided for 6 weeks.
  Interventions: Other: Tupler's Technique
- Control Group (Active Comparator): Traditional treatment protocol will be applied to this group that includes traditional exercises for diastasis rectus abdominis and this protocol will be followed 3 times per week for 6 weeks.
  Interventions: Other: Traditional Exercises

INTERVENTIONS:
Other: Tupler's Technique — Patient will wear diastasis rehab splint and will follow Tupler's techniqe protocol for 6 weeks. In the first 2 weeks both elevator and contracting exercises will be performed and after 2 weeks in the 3rd week only contracting exercises will be perform and for these exercises we divide abdomen into 6 floors and will patient have to contract her tummy towards the 3rd to 5th floor in first week, towards the 4th to 5th floor in 2nd week and from 5th to 6th floor in the 3rd week. in the wek 4 to week 6 head lifts will also be started along with contracting exercises from 5th to 6th floor.
  Arms: Interventional Group
Other: Traditional Exercises — The traditional treatment includes traditional abdominal exercises that patient will be perform for 6 weeks and three times per week with 15 repetitions of each exercise. These exercises includes posterior pelvic tilt' static abdominal contractions', reverse sit up exercise, kegals, russian twist , trunk twist and reverse trunk twist.
  Arms: Control Group

SUMMARY:
Diastasis Rectus Abdominis is the condition in which two abdominal muscles rectus abdominis separated and cause widening and thinning of Linea alba. The Tupler's Technique is Evidence Based intervention for the management of Diastasis Rectus Abdominis. The purpose of this study is to see the Effectiveness of Tupler's Technique on the Management of Diastasis Rectus Abdomins in Post-Partum Females.

DETAILED DESCRIPTION:
Literature suggest that during pregnancy due to hormonal changes such as increased in Relaxin, estrogen and progesterone level and also increased in the size of uterus affect the aponeurosis connection of abdominal muscles and due to these changes Diastasis Rectus Abdominis is common during pregnancy especially in third trimester and in the post-partum period. we can measure diastasis rectus abdominis by different methods such as palpatory, caliper and ultrasound. The condition can be mild (two fingers gap), moderate (two to three fingers gap) and severe (more than three fingers gap). The separation of greater than 2cm is considered as Diastasis Rectus Abdominis.

In this study effectiveness of Tupler's Technique will be assessed in post-partum diastasis rectus abdominis patients. Patients will have to wear diastasis rehab splints and then perform tupler's technique exercises. The mechanism behind this is when patients wear splint the splint will keep the connective tissues in narrow position for better healing and strengthening of muscles will be done by Tuper's Technique exercises and Diastasis of Rectus Abdominis willl be treated.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous and multiparous females (Vaginal delivery).
* Greater than and equal to 12 weeks post-partum
* Age limit will be18-30 years
* BMI under or equa to 29kg/m2
* Visiting with the complain of low back pain
* Diastasis of rectus abdominis at the level of umbilicus with mild, moderate and severe condition.

Exclusion Criteria:

* Other musculoskeletal disease (disc prolapse and disc bulge)
* Trauma of bowel and bladder
* Heart and respiratory conditions including sneezing and excessive coughing
* Any pelvic floor, abdominal and spinal surgery

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Digital nylon caliper to measure inter-recti Distance | Before intervention, after 3 weeks and after 6 weeks.
  Digital nylon caliper is the valid and reliable instrument to measure the inter-recti distance and inter-recti distance will be measured at three levels. at the level of umbilicus, 4.5cm above umbilicus and 4.5cm below umbilicus.
Oswestry low bac pain disability Questionnaire | Before intervention, after 3 weeks and after 6 weeks.
  This is a valid tool to assess back pain and this questionnaire has 10 sections and we grade level of disability according to grading criteria. 0-4shows no disability, 5-14 shows mild disability, and 15-24 shows moderate disability, and 25-34 shows severe disability and grade 35-50 means completely disabled.
Numeric Pain rating scale | Before intervention, after 3 weeks and after 6 weeks.
  By using this scale we will measure the intensity of back pain. i scores pain from 0-10. 0 means no pain, 5 means moderate pain and 10 means severe pain.
Maternal post-partum quality of life instrument (MPQOL-I) | Before intervention, after 3 weeks and after 6 weeks.
  This questionnaire has 5 domains. psychological, reltion with family and friends, relation with spouse, socioeconomic and health related domain and we can assess every domain of female life.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Study Chair — Riphah International University, Islamabad, Pakistan; Aqsa Shahid, MSPT*, Principal Investigator — Riphah International University, Islamabad, Pakistan
Locations (2):
- Pakistan (2):
  - Allied Hospital Faisalabad, Faisalābad, Punjab Province
  - Madinah Teaching Hospital Faisalabad, Faisalābad, Punjab Province

IPD SHARING:
Plan to Share IPD: No